CLINICAL TRIAL: NCT05217745
Title: A Randomised Controlled Pilot Study to Test the Role of Medium- and Long-chain Triacylglycerols (MLCT) in Reversing the Phenotype of Non-alcoholic Steatohepatitis (NASH) Patients
Brief Title: MLCT Oil for Fatty Liver - PASS Trial
Acronym: PASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Wilmar International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/00618
Record Dates: First submitted 2021-09-09; First posted 2022-02-01 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2021-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): MLCT oil (provided through ready to eat meals and snacks)
  Interventions: Dietary Supplement: MLCT Oil
- Control (Placebo Comparator): Corn oil (provided through ready to eat meals and snacks)
  Interventions: Dietary Supplement: LCT Oil (Corn Oil)

INTERVENTIONS:
Dietary Supplement: MLCT Oil — 1st 12 weeks: frozen ready to eat meals prepared with the oil Last 12 weeks: own diet with provided snacks containing the oil
  Arms: Treatment
Dietary Supplement: LCT Oil (Corn Oil) — 1st 12 weeks: frozen ready to eat meals prepared with the oil Last 12 weeks: own diet with provided snacks containing the oil
  Arms: Control

SUMMARY:
The main objective of this randomised pilot study is to explore the relative efficacy of dietary MLCT oil versus LCT oil (corn oil) in augmenting therapy of overweight and obese NAFLD patients with at least a 1-stage reversal between F1 and F4.

DETAILED DESCRIPTION:
The hypothesis of the study will be that daily intake of MLCT oil is more effective than corn oil in improving either NAFLD or NASH phenotype, with a greater reduction in liver fibrosis stage of participants with NASH.

The single-centre trial is a 2-arm, randomized pilot study with stratification by BMI. Up to 30 participants with biopsy/imaging proven NAFLD / NASH would undergo blinded 1:1 allocation to either control or test group.

All participants would be offered biopsy, whereby a repeat liver biopsy would be undertaken at the end of the study (6 months) to investigate the efficacy of dietary MLCT versus corn oil in augmenting therapy of NASH.

Dietary counselling for the participants will be provided by NUH dietician on 6 weekly basis on how to adhere to the required dietary regimen. For the first 12 weeks, participants are to consume only the 3 provided RTE meals (breakfast, lunch and dinner), with additional fruits or low calories snacks to be advised by dietician. During the second 12-week experimental period, participants will follow strict dietary guideline under the recommendation of the NUH dietician and have oil-containing products [chocolate sauce / oatmeal biscuits] with 30 g of corn or MLCT oil per day.

During the 6 months, study participants would be followed up at 0, 3, 6, 9, 12, 18 and 24 weeks. During each of the follow up visit, the participant would have blood drawn, urine and stool collected as per study schedule.

ELIGIBILITY:
Inclusion Criteria:

* Between 21 to 65 years old;
* Body mass index (BMI) 23 kg/m2 or higher;
* NAFLD or NASH as determined by liver biopsies within last 2 years with fibrosis stage F1-F4; OR Presence of steatosis and fibrosis via Transient Elastography / MRI
* Participants willing and able to adhere to the prohibitions and restrictions specified in the protocol;
* Participants willing and able to adhere to the dietary prescription as in the study protocol;
* Participants willing and able to provide written informed consent.
* Participants able to read and write English, and own a smartphone with a data plan

Exclusion Criteria:

* Poorly controlled diabetes
* Poorly controlled hypertension
* Estimated glomerular filtration rate of less than 60 ml/min/1.73m2;
* Presence of active alcoholic liver disease, chronic viral hepatitis, drug-induced hepatitis; autoimmune hepatitis, and liver cancer;
* A history of Type 1 diabetes mellitus or previous admission for diabetic ketoacidosis;
* Recurrent urinary tract infection (2 or more over the past one year);
* Having any medical condition that would affect metabolism (i.e. Cushing syndrome, known active hyperthyroidism or hypothyroidism);
* Serious medical disease with likely life expectancy less than 5 years;
* Recently started on selected diabetes / hypertensive medications. Must be on stable doses.
* Ongoing eating disorder or significant weight loss or weight gain as defined by change of 5% or more within 12 weeks before screening visit;
* History of any malignancy within 5 years of screening;
* Women who are pregnant or plan to become pregnant;
* Taking alcohol above the limit recommended (i.e. consumed more than 10 g/day for women or 20 g/day for men);
* Participation in other clinical trial in the 30 days before randomization;
* Participants who cannot be followed up for at least 6 weeks (due to health situation or travel);
* Having allergies / intolerances to the ingredients in the prepared meals or oil-containing products of the study;
* Having chronic gastrointestinal disorders;
* Having taken antibiotics in the last 3 months;
* Participants with arthropathy, CVM, CVA disorder or any systemic disorder which render or when intervention may be dangerous.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Liver Fibrosis | 6 months
  Change in liver fibrosis through liver biopsy or imaging

SECONDARY OUTCOMES:
Body Weight | 6 months
  Change in body weight (kg)
Body fat composition | 6 months
  Change in body fat composition using MRI body profiler (%)
Blood pressure | 6 months
  Change in blood pressure using blood pressure monitor (mmHg)
Body circumferences | 6 months
  Change in waist and hip circumference using measuring tape (cm)
Blood lipid profile (HDL, LDL, Total cholesterol, Triglycerides) | 6 months
  Change in fasting blood lipid profile (mmol/L)
Fasting Insulin and Glucose | 6 months
  Change in fasting Insulin and Glucose (mmol/L)
Haemoglobin A1c | 6 months
  Change in HBA1c (mmol/mol)
Liver function panel (Albumin, Bilirubin, ALT, AST, ALP, LDH, GGT) | 6 months
  Change in Albumin (g/L), bilirubin (umol/L), ALT, AST, ALP, LDH, GGT (U/L)
Creatinine | 6 months
  Change in serum and urine creatinine (umol/L)
Beta-hydroxybutyrate | 6 months
  Change in beta-hydroxybutyrate (mmol/L)
C-peptide | 6 months
  Change in C-peptide (pmol/L)
Oral glucose tolerance test | 6 months
  Change in glucose level at 120hr timepoint (mmol/L)
C-reactive protein (CRP) | 6 months
  Change in CRP (mg/L)
Inflammatory markers - IL-6, IL-1, TNFalpha | 6 months
  Change in inflammatory markers - IL-6, IL-1, TNFalpha
Gut microflora composition | 6 months
  Change in gut microbiota using gut metagenomics profiling

CONTACTS AND LOCATIONS:
Overall Officials: Dan Yock Young, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided